CLINICAL TRIAL: NCT05174715
Title: Evaluation of Malnutrition in Patients Undergoing Major Abdominal Surgery Using GLIM Criteria and Comparing CT and BIA for Muscle Mass Measurement
Brief Title: Malnutrition Using GLIM Criteria and Comparing CT and BIA for Muscle Mass Measurement
Status: Completed | Type: Observational
Sponsor: Klinikum St. Georg gGmbH (Other)
Responsible Party: Principal Investigator, Maria Wobith, Principle Investigator, Klinikum St. Georg gGmbH
Other Study IDs: GLIMCTBIA
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Malnutrition
Keywords: malnutrition, sarcopenia, GLIM criteria
MeSH Terms: conditions — Malnutrition; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: BIA — nutritional status was evaluated using BIA

SUMMARY:
Evaluation of malnutrition with the help of the GLIM criteria. Muscle mass measurement, as recommended in the GLIM criteria was done with the help of abdominal CT scan and BIA. Both methods were compared and their association to the clinical outcome was assessed.

DETAILED DESCRIPTION:
We retrospectively analysed 260 patients undergoing major abdominal surgery between January 2017 and December 2019. Patients were prospectively screened and assessed for malnutrition with Nutritional Risk Score (NRS) and Subjective Global assessment (SGA). Body composition was analysed with CT scan and BIA within 30 days before surgery. GLIM criteria were retrospectively determined referring to the Fat free Mass from BIA (FFMBIA) and Muscle Mass from axial CT scan at lumbar level 3 (MMCT). The prevalence of GLIM - malnutrition according to BIA and CT was evaluated. Multivariate logistic regression analysis was used to determine association between malnutrition and outcome parameters. ROC-curves specified sensitivity and specificity of the different tools and areas under the curve were calculated.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years
* BIA and CT scan was available within 31 days before surgery
* patients undergoing major abdominal surgery for gastrointestinal cancer

Exclusion Criteria:

* patients who were not able to agree to the participation
* missing assessment of the nutritional status
* leck of quality of the CT scan

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing major abdominal surgery for gastrointestinal cancer
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
overall complications | 31 days POD
  all complications perioperatively including surgical side infections, anastomic leakage, sepsis

IPD SHARING:
Plan to Share IPD: No